CLINICAL TRIAL: NCT05005442
Title: A Phase 2, Open-label Study to Evaluate the Safety and Efficacy of MK-7684A (MK-7684 [Vibostolimab] With MK-3475 [Pembrolizumab] Coformulation) in Participants With Relapsed or Refractory Hematological Malignancies
Brief Title: A Study of Pembrolizumab/Vibostolimab (MK-7684A) in Relapsed/Refractory Hematological Malignancies (MK-7684A-004, KEYVIBE-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7684A-004; MK-7684A-004 (Other: MSD); KEYVIBE-004 (Other: MSD); 2021-001700-15 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab/vibostolimab coformulation (Experimental): Participants will receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
  Interventions: Biological: Pembrolizumab/vibostolimab coformulation

INTERVENTIONS:
Biological: Pembrolizumab/vibostolimab coformulation — Pembrolizumab 200 mg + vibostolimab 200 mg/20 mL vial IV infusion Q3W up to approximately 2 years.
  Other Names: MK7684A

SUMMARY:
The purpose of the study is to determine the safety and tolerability of pembrolizumab/vibostolimab (MK-7684A) in hematological malignancies. This study will also evaluate the overall response rate (ORR), the duration of response (DOR), and disease control rate (DCR) following administration of pembrolizumab/vibostolimab. In addition, this study will characterize pharmacokinetic (PK) profile of vibostolimab (MK-7684).

ELIGIBILITY:
Inclusion Criteria

- Have confirmed relapsed/refractory classic Hodgkins Lymphoma (cHL), Primary mediastinal B-cell lymphoma (PMBCL), Follicular Lymphoma (FL), Diffuse large B-cell lymphoma (DLBCL) or Non-Hodgkins Lymphoma (NHL), or multiple myeloma (MM).

For PMBCL, DLBCL, FL, and MM:

- Must be relapsed or refractory to CAR-T-cell therapy or unable to receive it.

For DLBCL and NHL:

- Must have exhausted or be ineligible for or intolerant to all treatments, which in the opinion of the investigator are standard of care for their disease.

For NHL:

- Participants with Mantle cell lymphoma (MCL) must have received prior Bruton's tyrosine kinase inhibitor therapy.

All participants:

* Have measurable disease.
* Have adequate organ function.
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before allocation.
* Must be able to provide newly obtained bone marrow biopsy or aspirate material for disease assessment.
* Female participants are eligible to participate if not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of non child-bearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle.

Exclusion Criteria

For DLBCL and NHL:

- Has lymphoplasmacytic lymphomas, Waldenstrom's macroglobulinemia, chronic lymphocytic leukemia (not associated with small lymphocytic lymphoma), Burkitt (-like) lymphoma, mature T cell and NK cell neoplasms, immunodeficiency associated lymphoproliferative neoplasms, or histiocytic and dendritic cell neoplasms.

For MM:

* Has oligo-secretory myeloma, plasma cell leukemia, smoldering multiple myeloma, or monoclonal gammopathy of undetermined significance.
* Has a history of primary amyloidosis, hyperviscosity or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Has known prior or current central nervous system (CNS) involvement.

For Epstein Barr virus (EBV) positive DLBCL:

- Associated with a solid organ transplant.

For all participants:

* A WOCBP who has a positive urine pregnancy test within 72 hours before study intervention allocation.
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention.
* Has a history of a second malignancy.
* Any PMBCL participants that require the use of urgent cytoreductive therapy.
* If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery before starting study intervention.
* Has received prior radiotherapy within 2 weeks of start of study intervention.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention.
* Has a known severe hypersensitivity to MK-7684A, vibostolimab or pembrolizumab and/or any of its excipients.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has an active infection requiring systemic therapy.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks before enrollment.
* Has dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and Hepatitis C (HCV) infection (anti-HCV Ab (+) and detectable HCV RNA) at study entry..
* Has had an allogenic hematopoietic stem cell/solid organ transplantation within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (65):
- United States (9):
  - City of Hope Comprehensive Cancer Center-Hematology ( Site 0024), Duarte, California
  - University of Colorado Anschutz Medical Campus-The Center for Cancer and Blood Disorders ( Site 0021, Aurora, Colorado
  - University of Chicago Medical Center ( Site 0005), Chicago, Illinois
  - Henry Ford Hospital ( Site 0003), Detroit, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0004), Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0023), New Brunswick, New Jersey
  - University of Texas MD Anderson Cancer Center ( Site 0014), Houston, Texas
  - Medical Oncology Associates, PS ( Site 0001), Spokane, Washington
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0016), Milwaukee, Wisconsin
- Brazil (2):
  - Instituto do Câncer e Transplante de Curitiba ( Site 0611), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0601), Natal, Rio Grande do Norte
- Canada (4):
  - BC Cancer Vancouver ( Site 0034), Vancouver, British Columbia
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0031), Toronto, Ontario
  - Jewish General Hospital ( Site 0032), Montreal, Quebec
  - McGill University Health Centre ( Site 0037), Montreal, Quebec
- Chile (2):
  - Instituto Nacional del Cancer ( Site 0626), Chile, Region M. de Santiago
  - FALP-UIDO ( Site 0623), Santiago, Region M. de Santiago
- Denmark (2):
  - Rigshospitalet-Hematology - CTU ( Site 0361), Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby-Blodsygdomme ( Site 0362), Aarhus, Central Jutland
- France (3):
  - Gustave Roussy-DITEP ( Site 0301), Villejuif, Paris
  - centre hospitalier lyon sud-Service Hématologie ( Site 0300), Pierre-Bénite, Rhone
  - Pitie Salpetriere University Hospital-Clinical haematology ( Site 0304), Paris
- Germany (6):
  - Universitätsklinikum Marburg ( Site 0333), Marburg, Hesse
  - Universitaetsklinikum Koeln-Klinik I für Innere Medizin ( Site 0321), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 0327), Essen, North Rhine-Westphalia
  - Klinikum Mutterhaus der Borromäerinnen-Innere Medizin I ( Site 0325), Trier, Rhineland-Palatinate
  - Universitätsklinikum Leipzig ( Site 0328), Leipzig, Saxony
  - Universitaetsklinikum Hamburg-Eppendorf-II. medical clinic ( Site 0332), Hamburg
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Központ-I.sz. Belgyógyászati Klinika Hematológia ( Site 0401), Pécs, Baranya
  - Országos Onkológiai Intézet-HEMATOLÓGIA ÉS LYMPHOMA OSZTÁLY KEMOTERÁPIA A ( Site 0405), Budapest, Pest County
  - Semmelweis University-Belgyógyászati és Hematológiai Klinika ( Site 0403), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Haematologia) ( Site 0402), Debrecen
- Israel (5):
  - Soroka Medical Center-Hematology Department ( Site 0523), Beersheba
  - Rambam Health Care Campus ( Site 0526), Haifa
  - Hadassah Medical Center ( Site 0522), Jerusalem
  - Sheba Medical Center-Hemato Oncology ( Site 0524), Ramat Gan
  - Sourasky Medical Center ( Site 0525), Tel Aviv
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli-ISTITUTO DI EMATOLOGIA ( Site 0383), Rome, Lazio
  - Azienda Ospedaliera Spedali Civili di Brescia-Hemathology ( Site 0400), Brescia, Lombardy
  - Ospedale San Raffaele-Unità Linfomi ( Site 0382), Milan, Lombardy
  - Policlinico S. Orsola- Malpighi-Istituto di Ematologia "L. e A. Seragnoli" ( Site 0381), Bologna
- Poland (4):
  - Uniwersytecki Szpital Kliniczny-Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku ( Site, Wrocaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Chłonnego ( S, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 0424), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0427), Gliwice, Silesian Voivodeship
- Russia (4):
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 0548), Ufa, Baskortostan, Respublika
  - Almazov National Medical Research Centre-Intensive care unit No. 10 for oncohematological patients (, Saint Petersburg, Leningradskaya Oblast'
  - Moscow City Clinical Hospital S.P. Botkin ( Site 0547), Moscow, Moscow
  - Russian Scientific Research Institute of Hematology and Blood Transfusion-Hematology ( Site 0542), Saint Petersburg, Sankt-Peterburg
- Spain (4):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 0442), L'Hospitalet Del Llobregat, Barcelona
  - Clinica Universidad de Navarra ( Site 0444), Pamplona, Navarre
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 0446), Madrid
  - Hospital Universitario de Salamanca-Hematology ( Site 0441), Salamanca
- Taiwan (2):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 0263), Kaohsiung Niao Sung Dist, Kaohsiung
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0262), Taoyuan District
- Turkey (Türkiye) (6):
  - Ege University Medicine of Faculty ( Site 0565), Bornova, İzmir
  - Ankara University Hospital Cebeci ( Site 0561), Ankara
  - Mega Medipol-Hematology ( Site 0567), Istanbul
  - Vehbi Koc Vakfi - Amerikan Hastanesi ( Site 0562), Istanbul
  - Dokuz Eylül Üniversitesi-Hematology ( Site 0563), Izmir
  - Ondokuz Mayıs Universitesi ( Site 0564), Samsun
- Ukraine (4):
  - Cherkasy Regional Oncology Dispensary ( Site 0593), Cherkassy, Cherkasy Oblast
  - National Cancer Institute ( Site 0585), Kyiv, Kyivska Oblast
  - Institute of Transfusion Medicine and Blood of the National Academy of Medical Sciences of Ukraine (, Lviv, Lviv Oblast
  - National Research Center for Radiation Medicine of National Academy of Medical Sciences of Ukraine (, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred ninety-two participants were allocated, 1 participant was allocated but did not receive treatment due to worsening of underlying disease. No participants were enrolled into Part 2 of the study (The study was closed with amendment 5 after the last subject completed 35 cycles of the first course of Part 1).
Groups:
- Cohort A Pembrolizumab/Vibostolimab Coformulation: Participants with classic Hodgkin's lymphoma (cHL) or primary mediastinal B-cell lymphoma (PMBCL) who are relapsed or refractory to at least 1 line of prior therapy (cHL) of at least 2 lines of prior therapies (PMBCL) received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- Cohort B Pembrolizumab/Vibostolimab Coformulation: Participants with cHL or PMBCL who are relapsed or refractory to at least 2 lines of prior therapies (cHL) of at least 3 lines of prior therapies (PMBCL) received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- Cohort C Pembrolizumab/Vibostolimab Coformulation: Participants with relapsed or refractory follicular lymphoma (FL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- Cohort D Pembrolizumab/Vibostolimab Coformulation: Participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- Cohort E Pembrolizumab/Vibostolimab Coformulation: Participants with relapsed or refractory multiple myeloma (MM) following at least 3 lines of therapy and have exhausted all approved lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- Cohort F Pembrolizumab/Vibostolimab Coformulation: Participants with relapsed or refractory non-Hodgkin's lymphoma (NHL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
Period: Overall Study
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Started | 42 | 42 | 20 | 30 | 25 | 33
Treated | 42 | 42 | 20 | 30 | 25 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 42 | 42 | 20 | 30 | 25 | 33
Not completed — Death | 14 | 10 | 8 | 22 | 13 | 15
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Sponsor decision | 26 | 26 | 10 | 5 | 9 | 12
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 3 | 0 | 5
Not completed — Site terminated by sponsor | 0 | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation | Total
Number analyzed (Participants) | 42 | 42 | 20 | 30 | 25 | 33 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (16.5) | 46.7 (17.6) | 63.6 (12.8) | 60.7 (12.7) | 64.4 (10.8) | 66.0 (14.4) | 55.1 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 8 | 15 | 15 | 13 | 85
  Male | 24 | 26 | 12 | 15 | 10 | 20 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 3 | 5 | 1 | 3 | 21
  Not Hispanic or Latino | 36 | 33 | 15 | 22 | 24 | 29 | 159
  Unknown or Not Reported | 0 | 6 | 2 | 3 | 0 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 1 | 3 | 1 | 10
  White | 38 | 35 | 20 | 27 | 20 | 29 | 169
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 0 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Dose-Limiting Toxicity (DLT)
Description: A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). Percentage of participants who experience a DLT per CTCAE 5.0 are reported.
Time Frame: Up to approximately 6 weeks
Population: All participants who received at least one dose of study intervention and that finished the DLT evaluation period without a DLT or experienced a DLT in the DLT evaluation period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 42 | 41 | 18 | 20 | 10 | 25
Percentage of Participants | 4.8 [0.8 to 14.2] | 2.4 [0.1 to 10.8] | 0.0 [0.0 to 14.6] | 5.0 [0.3 to 20.8] | 0.0 [0.0 to 23.8] | 8.0 [1.4 to 22.8]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants who experience an AE are reported.
Time Frame: Up to approximately 27 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 42 | 42 | 20 | 30 | 25 | 32
Percentage of Participants | 92.9 | 97.6 | 95.0 | 80.0 | 80.0 | 87.5

3. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants discontinued from the study treatment due to an AE are reported.
Time Frame: Up to approximately 24 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 42 | 42 | 20 | 30 | 25 | 32
Percentage of Participants | 19.0 | 4.8 | 15.0 | 13.3 | 4.0 | 12.5

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Lugano 2014 Classification (Cohorts A-D & F)
Description: ORR for Cohorts A-D and F was assessed based on the Lugano 2014 Classification. ORR is defined as the percentage of the participants who had complete response (CR) or partial response (PR) and was evaluated using computed tomography (CT) and positron emission tomography (PET)-CT. CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). ORR for Cohorts A-D and F is presented. Cohort E is presented separately.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and had ORR measured by Lugano 2014 Classification.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 42 | 42 | 20 | 30 | 0 | 32
Percentage of Participants | 64.3 [48.0 to 78.4] | 35.7 [21.6 to 52.0] | 15.0 [3.2 to 37.9] | 16.7 [5.6 to 34.7] |  | 18.8 [7.2 to 36.4]

5. Secondary Outcome: ORR as Assessed by the 2016 International Myeloma Working Group (IMWG) Response Criteria (Cohort E)
Description: ORR for Cohort E was measured by 2016 IMWG Response Criteria. ORR is defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum Mprotein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The ORR for Cohort E is presented. Cohorts A-D and F were presented in a previous outcome measure.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and had ORR measured by the 2016 IMWG Response Criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 0
Percentage of Participants |  |  |  |  | 0.0 [0.0 to 13.7] |

6. Secondary Outcome: Duration of Response (DOR) as Assessed by Lugano 2014 Classification (Cohorts A-D & F)
Description: For participants who demonstrate a confirmed complete response (CR) or partial response (PR), DOR is defined as the time from CR or PR to documented disease progression or death. Participants are assessed using computed tomography (CT) and positron emission tomography (PET)- CT and response was evaluated based on the Lugano 2014 Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters (SPD) for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR for Cohorts A-D and F are presented. Cohort E is presented separately.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and had a response measured by measured by Lugano 2014 Classification.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 27 | 15 | 3 | 5 | 0 | 6
Months | 5.4 [2.9 to 11.00] | 3.0 [2.8 to 10.2] | 2.8 [2.8 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [2.9 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |  | 3.4 [1.6 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

7. Secondary Outcome: DOR as Assessed by 2016 IMWG Response Criteria (Cohort E)
Description: DOR is defined as the time from CR or PR to documented disease progression or death. DOR for Cohort E was measured by the 2016 IMWG Response Criteria with response criteria defined as participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR). CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum Mprotein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The DOR for Cohort E is presented. Cohorts A-D and F were presented in a previous outcome measure.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and had a response measured by measured by 2016 IMWG Response Criteria. No participants met the pre-specified analysis criteria for DOR in Cohort E (i.e., no participants with a response) and therefore DOR is unavailable for Cohort E.
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Disease Control Rate (DCR) as Assessed by Lugano 2014 Classification (Cohorts A-D & F)
Description: DCR is % of participants who had tumor response per response criteria or have stable disease (SD) for ≥ 12 weeks before any evidence of progressive disease (PD). CR or PR were evaluated with CT and PET-CT. CR: complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. PR: partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. DCR for Cohorts A-D & F are presented. Cohort E is presented in a separate outcome measure.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and were evaluated using Lugano 2014 Classification.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 42 | 42 | 20 | 30 | 0 | 32
Percentage of Participants | 73.8 [58.0 to 86.1] | 59.5 [43.3 to 74.4] | 25.0 [8.7 to 49.1] | 16.7 [5.6 to 34.7] |  | 31.3 [16.1 to 50.0]

9. Secondary Outcome: DCR as Assessed by 2016 IMWG Response Criteria (Cohort E)
Description: DCR: percentage of participants who have achieved tumor response or have shown SD for at least 12 weeks before any evidence of PD per IMWG response criteria 2016. Response criteria are defined as participants with either a sCR, CR, VGPR, or PR. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=CR as above PLUS normal serum FLC assay ratio and absence of clonal cells in bone marrow; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum Mprotein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. SD = Not meeting criteria for CR, VGPR, PR, or PD. PD as defined by prespecified 2016 IMWG response criteria. DCR for Cohort E is presented. Cohorts A-D and F were presented in a previous outcome measure.
Time Frame: Up to approximately 37 months
Population: All participants who have received at least one dose of study intervention and were evaluated using 2016 IMWG Response Criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 0
Percentage of Participants |  |  |  |  | 16.0 [4.5 to 36.1] |

10. Secondary Outcome: Lowest Plasma Concentration (Ctrough) of Vibostolimab
Description: Ctrough is the lowest concentration reached by a drug before the next dose is administered. Blood samples collected predose were used to determine Ctrough of Vibostolimab.
Time Frame: Predose at Cycles 1, 3, 7, 11, 15, 19, 23, 27 and 31. Cycle = 3 weeks
Population: All participants who received at least one dose of intervention and had data for the corresponding cycle.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 35 | 40 | 18 | 18 | 25 | 25
ug/mL
  Cycle 1 | 8.06 [6.71 to 9.68] | 9.86 [8.22 to 11.8] | 10.0 [6.61 to 15.3] | 9.64 [7.24 to 12.9] | 9.86 [6.52 to 14.9] | 9.52 [6.95 to 13.0]
  Cycle 3: number analyzed (Participants) | 34 | 37 | 14 | 10 | 4 | 17
  Cycle 3 | 15.3 [12.4 to 18.8] | 17.0 [13.3 to 21.6] | 22.6 [13.5 to 38.0] | 14.5 [7.55 to 27.9] | 17.9 [5.07 to 63.3] | 20.2 [15.8 to 25.9]
  Cycle 7: number analyzed (Participants) | 26 | 27 | 3 | 3 | 0 | 5
  Cycle 7 | 21.0 [17.1 to 25.8] | 19.5 [14.9 to 25.5] | 38.1 [6.15 to 236] | 25.8 [5.19 to 129] |  | 22.1 [14.1 to 34.7]
  Cycle 11: number analyzed (Participants) | 14 | 13 | 2 | 2 | 0 | 0
  Cycle 11 | 22.6 [16.6 to 30.8] | 24.2 [16.3 to 35.8] | 28.9 [0.251 to 3330] | 40.7 [40.1 to 41.4] |  |
  Cycle 15: number analyzed (Participants) | 11 | 6 | 0 | 2 | 0 | 0
  Cycle 15 | 26.2 [17.0 to 40.6] | 25.6 [17.4 to 37.8] |  | 40.6 [7.65 to 216] |  |
  Cycle 19: number analyzed (Participants) | 6 | 6 | 0 | 2 | 0 | 0
  Cycle 19 | 34.8 [21.6 to 56.2] | 24.2 [13.8 to 42.6] |  | 31.1 [5.49 to 176] |  |
  Cycle 23: number analyzed (Participants) | 4 | 6 | 0 | 1 | 0 | 0
  Cycle 23 | 36.5 [24.2 to 55.2] | 24.8 [15.2 to 40.3] |  | 51.5 [NA to NA] — Confidence interval cannot be calculated when N=1. |  |
  Cycle 27: number analyzed (Participants) | 4 | 4 | 0 | 2 | 0 | 0
  Cycle 27 | 40.6 [22.8 to 72.4] | 19.3 [9.23 to 40.4] |  | 48.9 [8.42 to 284] |  |
  Cycle 31: number analyzed (Participants) | 2 | 3 | 0 | 2 | 0 | 0
  Cycle 31 | 31.7 [2.43 to 413] | 31.6 [6.13 to 163] |  | 38.0 [1.57 to 923] |  |

11. Secondary Outcome: Maximum Concentration (Cmax) of Vibostolimab
Description: Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected post dose were used to determine Cmax of Vibostolimab.
Time Frame: Postdose: after end of infusion (up to ~10 minutes) at Cycles 1 and 8. Cycle = 3 weeks
Population: All participants who received at least one dose of intervention and had data for the corresponding cycle.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Cohort A Pembrolizumab/Vibostolimab Coformulation | Cohort B Pembrolizumab/Vibostolimab Coformulation | Cohort C Pembrolizumab/Vibostolimab Coformulation | Cohort D Pembrolizumab/Vibostolimab Coformulation | Cohort E Pembrolizumab/Vibostolimab Coformulation | Cohort F Pembrolizumab/Vibostolimab Coformulation
Number analyzed (Participants) | 37 | 38 | 17 | 26 | 24 | 28
ug/mL
  Cycle 1 | 85.8 [65.4 to 113] | 85.4 [70.0 to 104] | 42.6 [35.2 to 51.5] | 64.2 [54.2 to 76.1] | 53.2 [45.7 to 61.9] | 55.2 [44.2 to 69.0]
  Cycle 8: number analyzed (Participants) | 27 | 27 | 3 | 3 | 0 | 5
  Cycle 8 | 84.8 [69.9 to 103] | 75.8 [61.5 to 93.5] | 112 [22.8 to 552] | 77.4 [46.4 to 129] |  | 80.9 [58.4 to 112]

ADVERSE EVENTS:
Time Frame: Up to ~37 months.
Description: All-cause mortality: All allocated participants. Safety: All allocated participants who received at least 1 dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- COHORT A: Participants with classic Hodgkin's lymphoma (cHL) or primary mediastinal B-cell lymphoma (PMBCL) who are relapsed or refractory to at least 1 line of prior therapy (cHL) of at least 2 lines of prior therapies (PMBCL) received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- COHORT B: Participants with cHL or PMBCL who are relapsed or refractory to at least 2 lines of prior therapies (cHL) of at least 3 lines of prior therapies (PMBCL) received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- COHORT C: Participants with relapsed or refractory follicular lymphoma (FL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- COHORT D: Participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- COHORT E: Participants with relapsed or refractory multiple myeloma (MM) following at least 3 lines of therapy and have exhausted all approved lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
- COHORT F: Participants with relapsed or refractory non-Hodgkin's lymphoma (NHL) following at least 2 lines of therapy received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years.
Arm/Group | COHORT A | COHORT B | COHORT C | COHORT D | COHORT E | COHORT F
All-Cause Mortality (participants affected / at risk) | 14/42 | 10/42 | 9/20 | 24/30 | 14/25 | 15/33
Serious Adverse Events (participants affected / at risk) | 17/42 | 11/42 | 8/20 | 11/30 | 8/25 | 13/32
Other Adverse Events (participants affected / at risk) | 35/42 | 39/42 | 15/20 | 21/30 | 16/25 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT A (N=42) | COHORT B (N=42) | COHORT C (N=20) | COHORT D (N=30) | COHORT E (N=25) | COHORT F (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute cardiac event (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leydig cell tumour of the testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT A (N=42) | COHORT B (N=42) | COHORT C (N=20) | COHORT D (N=30) | COHORT E (N=25) | COHORT F (N=32)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 5 (6) | 1 (1) | 5 (5) | 7 (8) | 4 (5)
Eosinophilia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 8 (13) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (5) | 0 (0) | 4 (4) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 6 (6) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Hyperthermia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 7 (10) | 0 (0) | 4 (8) | 3 (4) | 4 (6)
COVID-19 (Infections and infestations) | 4 (4) | 7 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 3 (3) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 3 (3) | 0 (0) | 2 (4) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14) | 8 (13) | 1 (1) | 2 (2) | 1 (1) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05005442/Prot_SAP_000.pdf